CLINICAL TRIAL: NCT04019067
Title: Magnetically Controlled Capsule Endoscopy First vs. Standard Algorithm in Patients With Melena (FIRM Trial): a Multicenter, Randomized Controlled Trial
Brief Title: Magnetically Controlled Capsule Endoscopy First vs. Standard Algorithm in Patients With Melena
Acronym: FIRM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: few patients met all the inclusion criteria
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhuan Liao, M.D., Associate Professor, Associate Chief Physician, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MCE-melena-2019
Record Dates: First submitted 2019-07-12; First posted 2019-07-15 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Melena
Keywords: magnetically controlled capsule endoscopy; detection algorithm
MeSH Terms: conditions — Melena

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MCE first group (Experimental): Patients randomized to the "MCE first group" will have a MCE deployed as the first detection method.
  Interventions: Diagnostic Test: MCE first
- standard of care group (No Intervention): For patients randomized to the Standard Care Group, gastroenterologists choose which procedures to perform and when to perform them based on their interpretation of the patient's presentation.

INTERVENTIONS:
Diagnostic Test: MCE first — Patients randomized to the "MCE first group" will have a MCE deployed as soon as possible once confirmed to fast for at least 8 hours.
  Arms: MCE first group

SUMMARY:
MCE first algorithm is not inferior to standard of care algorithm in terms of further bleeding in hemodynamically stable patients with acute overt and non-hematochezia GI bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Presenting to the outpatient department or emergency department with melena (without hematemesis) within the previous 48 hours
* Hemodynamically stable (blood pressure > 100/60 mmHg and heart rate < 100 bpm) at presentation
* No endoscopy performed after the new onset of melena

Exclusion Criteria:

* Presenting with hematochezia and/or hematemesis within the previous 48 hours of presentation
* Hemodynamically stable after initial volume resuscitation
* Drop of hemoglobin level ≥ 2 g/dL/day, and/or need of transfusion ≥ 2 units of packed red blood cells per day
* Contraindications of CE (e.g. dysphagia, Zenker's diverticulum, esophageal stricture, known or suspected gastric or small bowel obstruction or perforation, gastroparesis, history of upper gastrointestinal surgery or abdominal surgery altering gastrointestinal anatomy, or post-abdominal radiation, etc.)
* Presence of internal cardiac defibrillator (ICD), pacemaker and/or other implanted electronic devices (cochlea, drug infusion pump, nerve stimulator, etc.) or magnetic metal foreign bodies; possibility of requiring an MRI examination prior to capsule excretion
* Patients who cannot undergo surgery in the event of capsule retention
* Pregnant and/or lactating women
* Patients with altered mental status (such as hepatic encephalopathy)
* Patients moribund from terminal malignant diseases or other end-stage illnesses with a limited life expectancy
* Unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
The rate of bleeding lesions detection. | 1 month
  Detection rate of bleeding lesions is defined as proportion of patients in whom a potential bleeding lesion is identified. Visualization of gross blood (fresh/coffee grounds) without any lesion will not be considered as a positive diagnosis. The panel will provide a diagnosis based upon the lesion presenting the highest potential for bleeding if there are many lesions detected.

SECONDARY OUTCOMES:
The time of the bleeding lesions detected from admission | 1 month
The number of procedures patients underwent for detection of the bleeding lesions | 1 month
The number of colonoscopy needed | 1 month
Rate of therapeutic intervention required of all patients | 1 month
  Therapeutic interventions include therapeutic endoscopy, radiologic intervention or surgery.
The length of hospital stay | 1 month
The cumulative direct cost of hospitalization | 1 month
Time to therapeutic intervention from presentation | 1 month
The rate of recurrent bleeding within 30 days of discharge | 1 month
  Further bleeding is defined as overt (hematemesis, melena or hematochezia) or occult (anemia or fecal occult blood positive) bleeding requiring subsequent hospitalization or transfusion, and/or signs of hypovolemic shock (systolic blood pressure of <100 mmHg and pulse rate >100 per min) or a drop-in hemoglobin level of >2g/dL per 24hours.
The all-cause mortality within 30 days of discharge | 1 month
Transfusion rate | 1 month

IPD SHARING:
Plan to Share IPD: No